CLINICAL TRIAL: NCT02247739
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, 3-Period Crossover Study to Evaluate the Efficacy and Safety of Recombinant Human C1 Inhibitor in the Prophylaxis of Angioedema Attacks in Patients With Hereditary Angioedema (HAE)
Brief Title: A Phase 2 HAE Prophylaxis Study With Recombinant Human C1 Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C1 3201
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Hereditary Angioedema
Keywords: HAE; Hereditary Angioedema; Prophylaxis
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; conestat alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- rhC1INH twice weekly (Experimental): rhC1INH administered twice weekly
  Interventions: Biological: Recombinant human C1 inhibitor
- rhC1INH once weekly (Experimental): rhC1INH administered once weekly
  Interventions: Biological: Recombinant human C1 inhibitor
- Placebo (Saline) twice weekly (Placebo Comparator): Placebo (Saline) administered twice weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Recombinant human C1 inhibitor
  Other Names: rhC1INH; Ruconest; Conestat alfa
  Arms: rhC1INH once weekly; rhC1INH twice weekly
Other: Placebo
  Other Names: Saline
  Arms: Placebo (Saline) twice weekly

SUMMARY:
Primary Objective:

To evaluate the efficacy of recombinant human C1 inhibitor (rhC1INH) in the prophylaxis of angioedema attacks in patients with HAE

Secondary Objective:

To evaluate the safety and immunogenicity of recombinant human C1 inhibitor (rhC1INH) in the prophylaxis of angioedema attacks in patients with HAE

DETAILED DESCRIPTION:
Study Design:

This is a multi-center, randomized, double-blind, placebo-controlled, 3-period crossover study of rhC1INH in prophylaxis of angioedema attacks in patients with HAE.

Medical screening (clinical and laboratory parameters) will be performed and patient medical history specific to HAE attacks will be collected to assess eligibility. Each patient will receive three 4 week periods of treatment twice weekly.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the following criteria at Screening are eligible for participation in the study:

1. Age 13 years or older
2. Laboratory confirmed diagnosis of HAE
3. A history of frequent HAE attacks (at least 4 attacks per month across a minimum of 3 consecutive months).
4. Female patients of childbearing potential who are sexually active must be willing to use an acceptable form of contraception.
5. Provided written informed consent (and written assent for minors)
6. Willingness and ability to comply with all protocol procedures

Exclusion Criteria:

Patients who meet any of the following criteria at Screening are to be excluded from study participation:

1. Patients with medical history of allergy to rabbits or rabbit-derived products (including rhC1INH)
2. Diagnosis of acquired angioedema (AAE)
3. Patients who are pregnant, or breastfeeding, or are currently intending to become pregnant
4. Treatment with any investigational drug in the past 30 days
5. Patients with any condition or treatment that, in the opinion of the Investigator, might interfere with the evaluation of study objectives
6. Patients currently treated with angiotensin-converting enzyme (ACE) inhibitors

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - University of South Florida Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - University of South Florida, Asthma, Allergy & Immunology Clinical Research Unit, Tampa, Florida
  - Washington University Division of Allergy and Immunology, St Louis, Missouri
  - Baker Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
- Ottawa Allergy Research Corp, Ottawa, Ontario, Canada
- Faculty Hospital by St. Anna Brno, Department of clinical Immunology and Allergology, Brno, Czechia
- Azienda Ospedaliera Universitaria Luigi Sacco Di Milano, Milan, Italy
- PHI University Clinic of Dermatology, Skopje, North Macedonia
- SC Centrul Clinic Mediquest SRL, Sângeorgiu de Mureş, Mureș County, Romania
- Clinical Center Serbia, Belgrade, Serbia

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Riedl MA, Grivcheva-Panovska V, Moldovan D, Baker J, Yang WH, Giannetti BM, Reshef A, Andrejevic S, Lockey RF, Hakl R, Kivity S, Harper JR, Relan A, Cicardi M. Recombinant human C1 esterase inhibitor for prophylaxis of hereditary angio-oedema: a phase 2, multicentre, randomised, double-blind, placebo-controlled crossover trial. Lancet. 2017 Sep 30;390(10102):1595-1602. doi: 10.1016/S0140-6736(17)31963-3. Epub 2017 Jul 25. PMID 28754491

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: rhC1INH twice weekly / rhC1INH once weekly / saline
- Treatments Sequence B: rhC1INH once weekly / rhC1INH twice weekly / Saline
- Treatment Sequesce C: Saline / rhC1INH once weekly / rhC1INH twice weekly
- Treatment Sequence D: Saline / rhC1INH twice weekly / rhC1INH once weekly
- Treatment Sequence E: rhC1INH twice weekly / saline / rhC1INH once weekly
- Treatment Sequence F: rhC1INH once weekly / saline / rhC1INH twice weekly
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatments Sequence B | Treatment Sequesce C | Treatment Sequence D | Treatment Sequence E | Treatment Sequence F
Started | 5 | 6 | 5 | 5 | 6 | 5
Completed | 5 | 3 | 4 | 5 | 5 | 4
Not Completed | 0 | 3 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Population is intention to treat (ITT) population
Groups:
- All Study Participants: All randomized patients
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 28
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 46 [17 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 2
  Czech Republic | 2
  Romania | 6
  United States | 7
  Macedonia, The Former Yugoslav Republic of | 8
  Italy | 1
  Serbia | 2
  Israel | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of HAE Attacks
Description: Average number of HAE attacks normalized to a 28 day period
Time Frame: 28 days
Population: Intent-to-Treat (ITT) Population: All patients who were randomized into one of the treatment sequences. The statistical analyses are based on the treatments to which the patient was randomized to receive during that treatment period.
Measure: Mean (95% Confidence Interval); unit: attacks
Groups:
- rhC1INH Twice Weekly: rhC1INH administered twice weekly
  Recombinant human C1 inhibitor
- rhC1INH Once Weekly: rhC1INH administered once weekly
  Recombinant human C1 inhibitor
- Placebo (Saline) Twice Weekly: Placebo (Saline) administered twice weekly
  Placebo
Arm/Group | rhC1INH Twice Weekly | rhC1INH Once Weekly | Placebo (Saline) Twice Weekly
Number analyzed (Participants) | 32 | 32 | 32
attacks | 2.74 [1.8 to 3.7] | 4.36 [3.1 to 5.6] | 7.18 [5.8 to 8.6]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants that experienced Treatment Emergent Adverse Events observed in safety population
Time Frame: 20 weeks
Population: Safety Population: All patients who received at least a partial injection of study drug. The statistical analyses are based on the actual treatment the patient received.
Measure: Count of Participants; unit: Participants
Arm/Group | rhC1INH Twice Weekly | rhC1INH Once Weekly | Placebo (Saline) Twice Weekly
Number analyzed (Participants) | 29 | 29 | 28
Participants | 10 | 13 | 8

3. Secondary Outcome: Percentage of Participants Achieving at Least 50% Reduction in Number of Attacks
Description: Percentage of participants achieving at least 50% reduction in the number of attacks normalized to a 28-day period as compared to the placebo treatment period
Time Frame: 28 days
Population: Both the rhC1INH twice weekly treatments and the rhC1INH once weekly treatment periods are compared to the placebo treatment for the safety population. One subject withdrew before receiving any treatment and is excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rhC1INH Twice Weekly | rhC1INH Once Weekly
Number analyzed (Participants) | 31 | 31
percentage of participants | 74 [57 to 86] | 42 [26 to 59]

4. Other Pre Specified Outcome: Immunogenicity
Description: Number of participants analyzed for neutralizing C1INH-specific antibodies and neutralizing rhC1INH-specific antibodies after confirmed anti-C1INH and anti rhC1INH IgM or IgG antibodies
Time Frame: 20 weeks
Population: Participants analyzed for Neutralizing antibodies after confirmed testing of anti-C1INH and anti rhC1INH IgM or IgG antibodies. Count of participants displays the number of positives.
Measure: Count of Participants; unit: Participants
Arm/Group | rhC1INH Twice Weekly | rhC1INH Once Weekly | Placebo (Saline) Twice Weekly
Number analyzed (Participants) | 3 | 5 | 2
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | rhC1INH Twice Weekly | rhC1INH Once Weekly | Placebo (Saline) Twice Weekly
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 5/29 | 7/29 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhC1INH Twice Weekly (N=29) | rhC1INH Once Weekly (N=29) | Placebo (Saline) Twice Weekly (N=28)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhC1INH Twice Weekly (N=29) | rhC1INH Once Weekly (N=29) | Placebo (Saline) Twice Weekly (N=28)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less